CLINICAL TRIAL: NCT07049640
Title: Acupressure and Cold Application on Pain, Anxiety, Comfort, and Hemodynamic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, Hediye Utli, PhD, RN, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: hediye1
Record Dates: First submitted 2025-06-18; First posted 2025-07-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Acupressure; Cold Application
Keywords: Pain; Anxiety; Comfort; Hemodynamic Parameters
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Acupressure Group Cold Application to Acupressure Points Group Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Experimental): Acupressure
  Interventions: Other: Acupressure Group
- Cold Application to Acupressure Points group (Active Comparator): Cold Application to Acupressure
  Interventions: Other: Cold Application to Acupressure Points Group
- Control group (No Intervention): Control

INTERVENTIONS:
Other: Acupressure Group — Effects of Acupressure Interventions
  Arms: Acupressure group
Other: Cold Application to Acupressure Points Group — Effects of Cold Application to Acupressure Points Interventions
  Arms: Cold Application to Acupressure Points group

SUMMARY:
The ventrogluteal injection is an invasive and often painful procedure commonly performed in healthcare settings. This study aimed to compare the effects of acupressure and cold application on pain, anxiety, comfort, and hemodynamic parameters prior to the ventrogluteal injection procedure.

Research questions

1. What is the effect of acupressure and cold application to acupressure points on pain caused by the ventrogluteal injection procedure?
2. What is the effect of acupressure and cold application to acupressure points on anxiety caused by the ventrogluteal injection procedure?
3. What is the effect of acupressure and cold application to acupressure points on comfort during the ventrogluteal injection procedure?
4. What is the effect of acupressure and cold application to acupressure points on pulse rate during the ventrogluteal injection procedure?
5. What is the effect of acupressure and cold application to acupressure points on respiratory rate during the ventrogluteal injection procedure?
6. What is the effect of acupressure and cold application to acupressure points on diastolic blood pressure during the ventrogluteal injection procedure?
7. What is the effect of acupressure and cold application to acupressure points on systolic blood pressure during the ventrogluteal injection procedure?

DETAILED DESCRIPTION:
Acupressure and cold application can significantly reduce pain associated with intramuscular injections. This simple, cost-effective, and easily applicable intervention can be utilized across various healthcare settings to alleviate injection-related discomfort.The aim of this study was to compare the effects of acupressure and cold application on pain, anxiety, comfort, and hemodynamic parameters prior to the ventrogluteal injection procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* Patients prescribed at least two doses of penicillin per day,
* There is an indication for injection administration
* Volunteer to participate in the research will be included.

Exclusion Criteria:

* Volunteer to participate in the research will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
NPR-Pain Scale | "Average of 3 months"
  The number 0 on the scale means they feel no pain or anxiety, while the number 10 represents the worst pain and the highest level of anxiety.
NPR-Anxiety Scale | "Average of 3 months"
  The number 0 on the scale means they feel no pain or anxiety, while the number 10 represents the worst pain and the highest level of anxiety.
Comfort Scale for Injection | "Average of 3 months"
  The lowest score that can be obtained from the scale is 1, and the highest score is 5.
Vital Signs follow-up Form | "Average of 3 months"
  Systolic and Diastolic Pressure 140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: HEDİYE ÖZBAY, PhD, Principal Investigator — Mardin Artuklu University
Locations (1):
- Siirt Training and Research Hospital, Siirt, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No